CLINICAL TRIAL: NCT00335322
Title: A Randomised, Open-label, 96-week Study Comparing the Safety and Efficacy of Three Different Combination Antiretroviral Regimens as Initial Therapy for HIV Infection.
Brief Title: ALTAIR - Alternative Antiretroviral Strategies : a Comparison of Three Initial Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCHECR-ALTAIR
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; efavirenz; Atazanavir Sulfate; Zidovudine; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Truvada (fixed dose combination of tenofovir + emtricitabine) + Stocrin efavirenz)
  Interventions: Drug: Truvada (fixed dose combination of tenofovir + emtricitabine) + Stocrin (efavirenz)
- 2 (Active Comparator): Truvada (fixed dose combination of tenofovir + emtricitabine)+ ritonavir/atazanavir (r/ATV)
  Interventions: Drug: Truvada (fixed dose combination of tenofovir + emtricitabine)+ ritonavir/atazanavir (r/ATV)
- 3 (Experimental): Truvada (fixed dose combination of tenofovir + emtricitabine) + zidovudine (ZDV) + abacavir (ABC)
  Interventions: Drug: Truvada (fixed dose combination of tenofovir + emtricitabine) + zidovudine (ZDV) + abacavir (ABC)

INTERVENTIONS:
Drug: Truvada (fixed dose combination of tenofovir + emtricitabine) + Stocrin (efavirenz) — Truvada (tenofovir 300mg qd + 200mg qd) once daily Efavirenz 600mg qd once daily
  Arms: 1
Drug: Truvada (fixed dose combination of tenofovir + emtricitabine)+ ritonavir/atazanavir (r/ATV) — Tuvada (tenofovir 300mg qd + 200mg qd) once daily ritoanvir/atazanavir 100mg/300mg qd once daily (taken with food)
  Arms: 2
Drug: Truvada (fixed dose combination of tenofovir + emtricitabine) + zidovudine (ZDV) + abacavir (ABC) — Tuvada (tenofovir 300mg qd + 200mg qd) once daily zidovudine 250mg/300mg qd (taken in two equal doses approximately 12 hours apart) Abacavir 600mg qd
  Arms: 3

SUMMARY:
In treatment naïve HIV infected subjects, combination antiretroviral therapy including efavirenz combined with tenofovir and emtricitabine will offer non-inferior antiretroviral efficacy over 48 weeks, compared to either atazanavir boosted with ritonavir combined with tenofovir and emtricitabine or tenofovir and emtricitabine combined with zidovudine and abacavir, as assessed by change from baseline plasma HIV-1 RNA viral load.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the virological efficacy, as measured by the time-weighted mean change from baseline plasma HIV-RNA, and safety, of three strategic regimens of initial antiretroviral therapy (ART) containing a fixed dose formulation of tenofovir and emtricitabine, with either efavirenz or ritonavir boosted atazanavir or zidovudine plus abacavir. (Primary comparisons are regimen I versus II and I versus III as described below).

I. tenofovir (TDF) + emtricitabine (FTC) + efavirenz (EFV) II. tenofovir (TDF) + emtricitabine (FTC) + ritonavir/atazanavir (r/ATV) III. tenofovir (TDF) + emtricitabine (FTC) + zidovudine (ZDV) + abacavir (ABC)

Secondary objectives of this study will be to undertake a range of analyses including but not limited to the following,

1. Percentage of patients < 50 copies HIV RNA/mL (and < 400 copies/mL) at week 48 and week 96 between treatment arms.
2. Time to confirmed (first of two consecutive) plasma HIV-1 RNA < 50 copies/mL (and < 400 copies/mL) between treatment arms.
3. Time to virologic failure defined as confirmed plasma HIV-1 RNA > 50 copies/mL (and 400 copies/mL) after confirmed < 50 copies/mL (where time = 0 if patient never achieves plasma virus load < 50 or <400 copies/mL).
4. Mean change from baseline of absolute CD4+ T cell count at weeks 48 and 96 between treatment arms.
5. Time to change in randomly assigned therapy (all reasons individually and on aggregate) between treatment arms.
6. Time to first virologic failure (defined as #3 above) or cessation of randomly assigned antiretroviral therapy.
7. Mean change from baseline Lipodystrophy Case Definition score at weeks 48 and 96 between treatment arms.
8. Mean change from baseline in peripheral and central adipose tissue, as measured by CT and DEXA at weeks 48 and 96 between treatment arms.
9. Mean change from baseline in fasting lipid and glycemic parameters at weeks 48 and 96 between treatment arms.
10. Comparison of total number of patients with any serious adverse events (SAEs), and the cumulative incidence of SAEs, between treatment arms.
11. Comparison of total number of patients with any adverse events (AEs), and the cumulative incidence of AEs, associated with cessation of randomly assigned therapy between treatment arms.
12. Patterns of genotypic HIV resistance associated with virological treatment failure across treatment arms.
13. Describe aspects of immune reconstitution disease.
14. Adherence to therapy and associations with virologic outcomes between treatment arms.
15. Comparison of quality of life between treatment arms.

Following the result of the scheduled week 48 data analysis, the protocol steering committee amended the study protocol as follows:

* Patients on Arms I and II will remain on the current study drugs
* Patients on Arm III may be switched at the physician's discretion to either Arm I or II
* There will be a protocol amendment to include one extra follow up visit at week 144 for all patients, regardless of treatment arm or current treatment
* All patients are to be encouraged to stay on the study up to week 144, to maximize follow up on study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive by licensed diagnostic test with presumed duration of infection > 6 months from date of randomisation.
* Aged > 16 years of age (or minimum age as determined by local regulations or as legal requirements dictate).
* Antiretroviral treatment naïve.
* Qualifying plasma HIV RNA > 2,000 copies/mL and a CD4+ T cell count of ≥ 50 cells/µL.
* No evidence of harbouring a drug resistant HIV (based upon genotypic drug testing).
* Calculated creatinine clearance (CLCr) greater than or equal to 70 mL/min (Cockcroft-Gault formula).
* Able to provide written informed consent.

Exclusion Criteria:

* The following laboratory variables,

  * absolute neutrophil count (ANC) < 750 cells/µL
  * haemoglobin < 8.0 g/dL
  * platelet count < 50,000 cells/µL
  * serum AST, ALT > 5 x upper limit of normal (ULN)
  * serum bilirubin > 1.5 x ULN
* Pregnant or nursing mothers.
* Current use of human growth hormone, testosterone or other anabolic steroid.
* Current use of any prohibited medications as described in product specific information.
* Acute therapy for serious infection or other serious medical illness (in the judgement of the site Principal Investigator) requiring systemic treatment and/or hospitalisation.
* Patients with current alcohol or illicit substance use that in the opinion of the site Principal Investigator would conflict with any aspect of the conduct of the trial.
* Patients unlikely to be able to remain in follow-up for the protocol-defined period.
* Patients with known renal insufficiency.
* Patients with obstructive liver disease.
* Patients with intractable diarrhoea (six loose stools/day for at least seven consecutive days).
* History of acute or chronic pancreatitis.
* Presence of cardiomyopathy (due to any cause) or any significant cardiovascular disease, such as unstable ischemic heart disease.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2007-02; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, AO DSc MD FRACP FRCPA FRCP, Principal Investigator — Kirby Institute

REFERENCES:
- [Result] Puls RL, Srasuebkul P, Petoumenos K, Boesecke C, Duncombe C, Belloso WH, Molina JM, Li L, Avihingsanon A, Gazzard B, Cooper DA, Emery S; Altair Study Group. Efavirenz versus boosted atazanavir or zidovudine and abacavir in antiretroviral treatment-naive, HIV-infected subjects: week 48 data from the Altair study. Clin Infect Dis. 2010 Oct 1;51(7):855-64. doi: 10.1086/656363. PMID 20735258
- [Result] Winston A, Duncombe C, Li PC, Gill JM, Kerr SJ, Puls R, Petoumenos K, Taylor-Robinson SD, Emery S, Cooper DA; Altair Study Group. Does choice of combination antiretroviral therapy (cART) alter changes in cerebral function testing after 48 weeks in treatment-naive, HIV-1-infected individuals commencing cART? A randomized, controlled study. Clin Infect Dis. 2010 Mar 15;50(6):920-9. doi: 10.1086/650743. PMID 20146627
- [Derived] Berthon-Jones N, Courtney-Vega K, Donaldson A, Haskelberg H, Emery S, Puls R. Assessing site performance in the Altair study, a multinational clinical trial. Trials. 2015 Apr 8;16:138. doi: 10.1186/s13063-015-0653-x. PMID 25872747
- See also: The Kirby Institute homepage (formerly known as the National Centre in HIV Epidemiology and Clinical Research) — https://kirby.unsw.edu.au/

RESULTS

PARTICIPANT FLOW:
Groups:
- TDF/FTC+EFV: Truvada (fixed dose combination of tenofovir+emtricitabine) + Stocrin efavirenz
- TDF/FTC+r/ATV: Truvada (fixed dose combination of tenofovir + emtricitabine)+ ritonavir/atazanavir (r/ATV)
- TDF/FTC+AZT+ABC: Truvada (fixed dose combination of tenofovir + emtricitabine) + zidovudine (ZDV) + abacavir (ABC)
Period: Overall Study
Arm/Group | TDF/FTC+EFV | TDF/FTC+r/ATV | TDF/FTC+AZT+ABC
Started | 115 | 107 | 105
Completed | 114 | 105 | 103
Not Completed | 1 | 2 | 2
Not completed — Randomised but withdrew prior to ART sta | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- TDF/FTC+EFV: Truvada (fixed dose combination of tenofovir + emtricitabine)+ Stocrin efavirenz
- Total: Total of all reporting groups
Arm/Group | TDF/FTC+EFV | TDF/FTC+r/ATV | TDF/FTC+AZT+ABC | Total
Number analyzed (Participants) | 115 | 107 | 105 | 327
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 107 | 105 | 327
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 22 | 76
  Male | 91 | 77 | 83 | 251
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 35 | 37 | 35 | 107
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 7 | 10 | 27
  White | 46 | 43 | 35 | 124
  More than one race | 24 | 20 | 25 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Mean Change From Baseline Plasma HIV-RNA.
Time Frame: 48 weeks
Population: Modified ITT; all randomised pts who started drug
Measure: Mean (95% Confidence Interval); unit: log copies/mL
Groups:
- TDF/FTC+EFV: Truvada (fixed dose combination of tenofovir + emtricitabine) + Stocrin (efavirenz)
  Truvada (tenofovir 300mg qd + 200mg qd) once daily Efavirenz 600mg qd once daily
- TDF/FTC+r/ATV: Truvada (fixed dose combination of tenofovir + emtricitabine) + ritonavir/atazanavir (r/ATV)
  Truvada (tenofovir 300mg qd + 200mg qd) once daily Ritonavir/atazanavi 100mg/300mg qd once daily
- TDF/FTC+AZT+ABC: Truvada (fixed dose combination of tenofovir + emtricitabine) + zidovudine + abacavir
  Truvada (tenofovir 300mg qd + 200mg qd) once daily Zidovudine 250mg/300mg qd taken in two equal doses approx. 12 hours apart Abacavir 600mg qd
Arm/Group | TDF/FTC+EFV | TDF/FTC+r/ATV | TDF/FTC+AZT+ABC
Number analyzed (Participants) | 114 | 105 | 103
log copies/mL | -2.59 [-2.67 to -2.41] | -2.69 [-2.89 to -2.49] | -2.39 [-2.54 to -2.24]

2. Secondary Outcome: Time Weighted Mean Change From Baseline Plasma HIV-RNA
Time Frame: 144 weeks
Population: Intent to Treat
Measure: Mean (95% Confidence Interval); unit: log copies/mL
Groups:
- TDF/FTC+EFV: Truvada (fixed dose combination of tenofovir + emtricitabine) + Stocrin (efavirenz): Truvada (tenofovir 300mg qd + 200mg qd) once daily Efavirenz 600mg qd once daily
- TDF/FTC+ r/ATV: Truvada (fixed dose combination of tenofovir + emtricitabine)+ ritonavir/atazanavir (r/ATV): Tuvada (tenofovir 300mg qd + 200mg qd) once daily ritoanvir/atazanavir 100mg/300mg qd once daily (taken with food)
- TDF/FTC + AZT+ABC: Truvada (fixed dose combination of tenofovir + emtricitabine) + zidovudine (ZDV) + abacavir (ABC): Tuvada (tenofovir 300mg qd + 200mg qd) once daily zidovudine 250mg/300mg qd (taken in two equal doses approximately 12 hours apart) Abacavir 600mg qd
Arm/Group | TDF/FTC+EFV | TDF/FTC+ r/ATV | TDF/FTC + AZT+ABC
Number analyzed (Participants) | 114 | 105 | 103
log copies/mL | -2.77 [-2.89 to -2.65] | -2.88 [-2.99 to -2.78] | -2.54 [-2.72 to -2.37]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TDF/FTC+EFV | TDF/FTC+r/ATV | TDF/FTC+AZT+ABC
Serious Adverse Events (participants affected / at risk) | 14/115 | 8/105 | 12/103
Other Adverse Events (participants affected / at risk) | 99/115 | 95/105 | 91/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF/FTC+EFV (N=115) | TDF/FTC+r/ATV (N=105) | TDF/FTC+AZT+ABC (N=103)
Autoimmune disorder (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
decreased blood pressure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (3)
Fatal outcome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
General systems disorder (General disorders) | 0 (0) | 1 (2) | 2 (2)
infection class unspecified (Infections and infestations) | 3 (4) | 1 (1) | 2 (4)
injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Investigations, imaging and histopathology (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
maternal complications of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Ovarian and fallopian tube disorders (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Pleural disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Therapeutic procedure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular hemorrhagic disorders (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous varices (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Viral infectious disorder (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
cardiac arrhythmias (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (5)
Depressed mood and disturbance (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anemias and marrow depression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal motility and defaecation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic conditions (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Hematological and lymphoid tissue therapeutic procedures (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic and heaptobiliary disroders (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF/FTC+EFV (N=115) | TDF/FTC+r/ATV (N=105) | TDF/FTC+AZT+ABC (N=103)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 11 (11)
Allergic condition (Immune system disorders) | 11 (11) | 10 (10) | 5 (5)
Body temperature disorders (General disorders) | 13 (13) | 8 (8) | 6 (6)
Bacterial infections (Infections and infestations) | 4 (4) | 9 (9) | 11 (11)
Reduced blood pressure disorders (Blood and lymphatic system disorders) | 36 (36) | 4 (4) | 10 (10)
Depressed mood (Psychiatric disorders) | 7 (7) | 1 (1) | 4 (4)
Fungal infections (Infections and infestations) | 11 (11) | 6 (6) | 8 (8)
Gastrointestinal motility and defaecation disorders (Gastrointestinal disorders) | 21 (21) | 18 (18) | 16 (16)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 24 (24) | 33 (33) | 68 (68)
General systems disorder (General disorders) | 17 (17) | 15 (15) | 15 (15)
headaches (Nervous system disorders) | 11 (11) | 11 (11) | 12 (12)
heaptic and hepatobiliary disorders (Hepatobiliary disorders) | 4 (4) | 46 (46) | 1 (1)
Infections - pathogennot specified (Infections and infestations) | 45 (45) | 36 (36) | 32 (32)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 11 (11) | 8 (8) | 9 (9)
Respiratory disroder NEC (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 8 (8) | 15 (15)
Sleep disorders (Psychiatric disorders) | 33 (33) | 8 (8) | 10 (10)
Viral infections (Infections and infestations) | 17 (17) | 11 (11) | 19 (19)
Epidermal and dermal disorders (Skin and subcutaneous tissue disorders) | 29 (29) | 14 (14) | 14 (14)

LIMITATIONS AND CAVEATS:
Inadequate sample size for true comparison of non-inferiority

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes